Official Title: The Effects of Electrical Muscle Stimulation Exercise on Upper, Lower

Extremity and Core Strength in Sedentary Women

NCT Number: Pending

Date: October 7, 2025

Prepared by: Dr. Ali Kerim Yılmaz

Esra Korkmaz Salkılıç

Institution: 19 Mayıs University

# **INFORMED CONSENT FORM\***

# STUDY TITLE (FULL TITLE OF THE STUDY)

The Effect of Electrical Muscle Stimulation Exercise on Lower, Upper Extremity, and Core Strength in Sedentary Women

#### **Volunteer's Initials << >>**

You are being asked to participate in a research study. Before deciding whether to participate, it is important that you understand why the research is being conducted, how your information will be used, what the study involves, the potential benefits, risks, and any concerns you may have. Please take the time to read the information below carefully and, if you wish, discuss this with your doctor or family physician. You cannot take part in this study if you are participating in another study.

## **DO I HAVE TO PARTICIPATE IN THIS STUDY?**

The decision to participate in the study is entirely yours. If you decide to participate, you will be given this Informed Consent Form to sign. If you decide to participate, you are free to withdraw from the study at any time. This will not affect the standard of care you receive. Your physician/family doctor will be informed of your participation in this clinical trial if you so choose.

#### WHAT IS THE SUBJECT AND PURPOSE OF THE STUDY?

Investigation of the effects of electrical muscle stimulation exercise on lower, upper extremity and core region strength in sedentary women.

#### **WORKING PROCEDURES:**

Before the study, you, as a participant, will be thoroughly informed and included in the study. Participants will be asked to complete a total of 10 laboratory visits: four before the 8-week exercise program, and three after the 8-week exercise program. During the first visit, participants will be informed about the tests and their age, height, weight, and body mass index will be measured. Both groups will follow the same exercise protocol. Anthropometric measurements will then be taken, and a trial will be administered. During the pre-, mid-(Week 4), and post-test periods, participants will complete a total of nine visits, three at 24-hour intervals, based on the test protocols they selected from the application cards provided for each period. Mid- and post-tests will be scheduled to avoid training days. All measurements and exercises will be performed in the gym at the same time of day (12:00-16:00). The content and scope of the exercises are designed to impact lower, upper, and core strength. For each measurement, you will need to allocate approximately 1 hour of your time to the measurements.

#### **Applications:**

- 1. Modifiye push up Test
- 2. Handgrip Strength Test (HS)
- 3. Bent Arm Hanging Test (BAH)
- 4. Single Leg Hop Tests (SLHT)
- 5. Deep squat
- 6. V-Sit Fleksör Test
- 7. Sit- Up Test

# WHAT SHOULD I DO?

You must be willing to comply with your study doctor's instructions and participate in the testing protocols. You must perform at your fullest during the testing protocols. You must arrive prepared for the tests on the dates and times specified by your study doctor, wearing appropriate attire, and you must inquire about the next test date and time from your doctor. It is also important to inform your study doctor of any other medical treatment you are receiving before or during the study.

#### What possible side effects, risks, and discomforts are there in participating in the study?

What possible side effects, risks, and discomforts are there in participating in the study?

#### WHAT ARE THE POSSIBLE BENEFITS OF PARTICIPATING IN THE STUDY?

Participants in the EMS group may experience improvements in muscle strength across the upper extremity, lower extremity, and core regions, as well as reductions in certain anthropometric measurements such as waist, hip, and abdominal circumference. Compared to traditional exercise protocols, EMS-assisted training may offer enhanced muscle activation and metabolic efficiency in a shorter time frame. While individual results may vary, the study may contribute to improved physical performance, body composition, and functional fitness in sedentary women. All participants will also be provided with feedback on their performance assessments upon completion of the study.

#### **VOLUNTARY PARTICIPATION**

My decision to participate in this study is entirely voluntary. I am aware that I can refuse to participate in this study or withdraw at any time after participation, without any liability or impact on the care and treatment I receive at this institution. If I withdraw from the study at any time, I will discuss my reasons for withdrawal, the consequences of my withdrawal, and any subsequent treatments I may receive with my doctor.

#### WHAT IS THE COST OF PARTICIPATING IN THE STUDY?

All test equipment related to the study will be provided by the Yaşar Doğu Faculty of Sports Sciences performance laboratories and the Farivar Wellness Center, so there will be no cost. There will be no fee charged to you or your private insurance or official social security institution.

#### HOW WILL MY PERSONAL INFORMATION BE USED?

By signing this form, you consent to your doctor and their staff collecting and using your personal information ("Study Data") for the study. This includes your date of birth, gender, and ethnicity. There is no specific timeframe for the use of your study data. However, you can withdraw your consent at any time by informing your doctor.

Your doctor will use your study data for the study. The institution where your doctor works is responsible for managing your study data in accordance with applicable data protection laws.

The results of the study may be published in medical journals, but your identity will not be disclosed in these publications.

Your doctor has the right to request information about your collected study data. You also have the right to request correction of any errors in this data. If you have any requests regarding this matter, please contact your doctor if necessary.

If you withdraw your consent, your doctor will no longer be able to use your study data or share it with others.

By signing this form, I consent to the use of your study data as described in this form.

# PEOPLE WHO CAN BE REACHED 24 HOURS DURING THE RESEARCH:

Name Surname Phone

Dr. Öğr. Üyesi Ali Kerim YILMAZ 0542 495 37 37

Esra KORKMAZ 0555 895 81 97

## SITUATIONS THAT WILL REQUIRE ME TO LEAVE THE WORK:

There are no side effects from the measurements taken. However, if you experience any health problems or feel unwell during the measurements, you can withdraw from the study at any time.

#### HOW MAY NEW INFORMATION AFFECT MY ROLE IN THE STUDY

Any new information that emerges during the work will be communicated to me immediately.

### **Consent to Participate in the Study**

I have read all the information in the Informed Consent Form. The physician listed below provided me with both written and verbal explanations regarding the research, the subject and purpose of which are outlined above. I understand that I am participating in the research voluntarily, that I may withdraw from the research at any time, with or without justification, and that I may be excluded from the research by the researcher regardless of my wishes.

I agree to participate in this research voluntarily, without any pressure or coercion. My physician has provided me with a copy of this document for safekeeping, including the points to be considered during the study.

Volunteer's Name Surname : Signature:

Date:

| Person Making the Statements | Name Surname: |
|------------------------------|---------------|
| | Signature: |

Date:

If necessary, the person who witnessed the consent process

Name Surname:

Signature: Date :

Legal Representative if necessary Name Surname

Signature Date: